CLINICAL TRIAL: NCT02717975
Title: A Prospective, Multicenter, Randomized Trial: The Effect of Catheter Valve Vs. Standard Catheter Removal in Outpatient Settings on the Patient Discharge Timings
Brief Title: The Effect of Catheter Valve Vs. Standard Catheter Removal in Outpatients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Shikohe Masood, Consultant Urological Surgeon, Medway NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 191435
Record Dates: First submitted 2016-01-20; First posted 2016-03-24 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Urinary Retention
Keywords: Urinary retention; trial removal of catheter; valve
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without valve (Active Comparator): Trial removal of catheter without catheter valve in patients with urinary retention. These are those patients who have catheter on free drainage, attend the clinic for catheter removal and bladder to be filled naturally ( which may take upto 4-5 hours). After removal of catheter they will be asked to drink plenty of fluids while waiting for the bladder to fill up.
  This is the traditional method of catheter removal.
  Interventions: Procedure: Trial removal of catheter in patients with urinary retention
- With valve (Experimental): Trial removal of catheter in patients with urinary retention with closed catheter valve. These patients will be asked to close the valve 3-4 hours before attending the clinic prior to catheter removal. Here the intervention is catheter valve that allows bladder to be comfortably full by the time patient arrives in the clinic. By this intervention the investigators hypothesise that the investigators can save the clinic time as the patient will not need to wait for natural bladder filling which generally takes 4-5 hours.
  Intervention: Urinary catheter valve
  Interventions: Procedure: Use of catheter valve before 'trial removal of catheter'

INTERVENTIONS:
Procedure: Use of catheter valve before 'trial removal of catheter' — The investigators are comparing two groups of patients (Group A) Trial removal of urinary catheter in patients with urinary retention after applying catheter valve and closing it 3-4 hours before catheter removal.
  Arms: With valve
Procedure: Trial removal of catheter in patients with urinary retention — The investigators are comparing two groups of patients (Group B) Trial removal of urinary catheter in patients with urinary retention without using catheter valve - 'Traditional method'
  Arms: Without valve

SUMMARY:
It is estimated that over 10% of men above the age of 60 will experience an episode of urinary retention over a period of 5 years and will need urethral catheter. Some of these patients are discharged from the hospital with urethral catheter, for them to attend a Trial Without Catheter (TWOC) clinic at a later date for catheter removal. Traditionally after catheter is removed in the clinic the nurse has to wait for up to 5 hours before the patient get the urge to pass urine and empty the bladder.

The main objective of this study is to see the effect of catheter valve on the length of clinic stay (timing of discharge)for the patients (men age 60-85) after catheter is removed.

In this study after randomization, patients in Group A (catheter valve group) will be given a catheter valve before they are sent home with the catheter.They will be asked to close the valve 3-4 hours (time required for adequate filling of bladder, which means minimum of 250 mls in bladder with natural filling) before their appointment. It is very likely that by the time these patients are seen in the TWOC clinic their bladder is already full and they will void soon after removal of catheter.The patients in Group B (control) will go home with free drainage catheter and urine bag (standard catheter removal). These patients on arrival, in the TWOC clinic will have an empty bladder when their catheter is removed, they will then drink plenty of fluids in the clinic and wait for their bladder to be full before they void spontaneously.

This study will last for one year after approval by ethical committee.

The time saved in this process would lessen patient anxiety, lead to more patients being reviewed in clinic and therefore reduced waiting times in TWOC clinics and will save money.

DETAILED DESCRIPTION:
Men who are discharged from the hospital with urinary catheter in situ are given an appointment to come to trial TWOC (trail without catheter) clinic for removal of their catheters.

Purpose and design:

In the TWOC clinic their catheters are removed and they usually wait for up to 5 hours hours before they get an urge to pass urine and empty the bladder and then sent home by the nurse. Waiting for up to 5 hours in the clinic reduces patient satisfaction and increases their anxiety. It also keeps the urology nurse busy in the clinic. This is shown by a clinical audit, which has been carried out in our department.

The aim of this study is to find out the ways to reduce this waiting time for the patients. In this study catheter valve is used to see if it significantly reduces time spent by the patient in the TWOC clinic after catheter removal. The patients in the catheter valve group are compared to the patients who did not use the valve (this is the standard method which is currently used by most of the TWOC clinics).

Catheter valve is a device, which is attached to the end of urinary catheter and can be used easily by any one who has normal manual dexterity and no cognitive impairment.

The study proposal was developed by lead urology nurse practitioner and endorsed by the consultant urological surgeons from three different hospitals in Kent UK (Medway Maritime Hospital, Darent Valley Hospital and Maidstone Hospital).

Recruitment:

Patients will be identified and recruited in the hospital ward. The patients who are planned to go home with the catheter will be provided with the patient information leaflet about his study. They will be given 6 hours to decide if they want to participate in this study. Those patients who agree to participate will be asked to sign a written informed consent. A computer-generated randomisation will be carried out. They will be given a contact number of the urology nurse in case they have any problems or if they want to ask any questions before attending TWOC clinic.

A day after discharge urology nurse practitioner will ring the patient at home to check if the patient still wants to participate in this study. A day before their appointment for TWOC clinic urology nurse will ring the patient (in Group A, valve group) to remind him about the appointment and also remind him to close the valve 3-4 hours before appointment time and patients in both groups (Group A and Group B) to drink three glasses of water before coming to the hospital for catheter removal. Patients will be informed that they can withdraw from the study at any point.

Inclusion and exclusion:

A strict inclusion and exclusion criteria will be observed. Vulnerable men with learning difficulties/dementia/Alzheimer's disease or those with poor manual dexterity will not be included.

Consent:

Written informed consent will be used after patients has read the patient information leaflet and the study has been verbally explained to the patient by the researchers.

Risks, burdens and benefits

There is no potential risk to the patients associated with the planned intervention.The vulnerable adults with learning difficulties/Dementia and poor manual dexterity will be excluded. In the intervention arm (GROUP A: patient with valve) the patient may get a pain with strong desire to pass urine or start bypassing catheter much before 3 hours after closing the valve. In this case patients will be instructed to open the valve and drain the urine. (These patients will be excluded).

If there is significant reduction (one hour or more) in the time spent in the clinic for the valve group noted in this study that will help in decreasing patient's anxiety, improved efficacy of the TWOC clinic and reduce the cost of running the TWOC clinic.

Confidentiality:

The data will be recorded electronically and will be saved in a password protected computer. The researchers and statistician can only access it.

Conflict of interest:

There is no conflict of interest. All the researchers will sign the form.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 60-85 catheterised for urinary retention and booked for outpatient removal of catheter
* Mobile patients

Exclusion Criteria:

* Who cannot consent
* Residual urine of more then 1 litre
* Abnormal renal functions
* Poor manual dexterity
* Learning difficulties/dementia.

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Time to spontaneous void after catheter removal | On the day of catheter removal
  The primary outcome measure of this study is to see if usage of catheter valve results in early spontaneous voiding after catheter removal and thus significantly reduces the time spent by these patients in the clinic.

SECONDARY OUTCOMES:
Complications associated with valve | On the day of catheter removal
  To see if the patients with the catheter valve have more complications (catheter bypass, urinary tract infection and pain).
Reduction in clinic waiting time (hours) | On the day of catheter removal
  To see if usage of catheter valve results in early discharge after catheter removal resulting in reduction of time spent in the clinic (in hours)
Reduction in the cost of running the clinic | On the day of catheter removal
  To see if reduction in the time spent by the catheter valve patients results in reducing the cost of running of the TWOC (Trial without catheter) clinic (in British Pound Sterling).

CONTACTS AND LOCATIONS:
Overall Officials: Shikohe Masood, MD, Principal Investigator — Medway NHS Foundation Trust
Locations (1):
- Medway NHS Foundation Trust, Gillingham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacobsen SJ, Jacobson DJ, Girman CJ, Roberts RO, Rhodes T, Guess HA, Lieber MM. Natural history of prostatism: risk factors for acute urinary retention. J Urol. 1997 Aug;158(2):481-7. doi: 10.1016/s0022-5347(01)64508-7. PMID 9224329
- [Background] Lyth DR, Braslis K, Iacovou JW. The infusion trial of micturition. Br J Urol. 1997 Jan;79(1):94-5. doi: 10.1046/j.1464-410x.1997.30520.x. PMID 9043505
- [Background] Boccola MA, Sharma A, Taylor C, Wong LM, Travis D, Chan S. The infusion method trial of void vs standard catheter removal in the outpatient setting: a prospective randomized trial. BJU Int. 2011 Apr;107 Suppl 3:43-6. doi: 10.1111/j.1464-410X.2011.10044.x. PMID 21492377
- [Background] Du J, Marshall D, Leyland J, Shaw L, Broome KE, Mason DF. Prospective, multicentre, randomized controlled trial of bladder filling prior to trial of void on the timing of discharge. ANZ J Surg. 2013 Apr;83(4):239-42. doi: 10.1111/j.1445-2197.2012.06253.x. Epub 2012 Sep 18. PMID 22984818
- [Background] Wilson C, Sandhu SS, Kaisary AV. A prospective randomized study comparing a catheter-valve with a standard drainage system. Br J Urol. 1997 Dec;80(6):915-7. doi: 10.1046/j.1464-410x.1997.00473.x. PMID 9439409
- [Background] German K, Rowley P, Stone D, Kumar U, Blackford HN. A randomized cross-over study comparing the use of a catheter valve and a leg-bag in urethrally catheterized male patients. Br J Urol. 1997 Jan;79(1):96-8. doi: 10.1046/j.1464-410x.1997.30321.x. PMID 9043506